CLINICAL TRIAL: NCT06085651
Title: To Explore the Risk Factors of Postoperative Shoulder Imbalance After Selective Thoracolumbar Fusion (STLF) Surgery in Adolescent Idiopathic Scoliosis(AIS)
Brief Title: The Relaionship Between Sagittal Spinal Parameters and PSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-225
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis; postoperative shoulder imbalance
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSI group: we divided all patients into two groups according to their RSH in the final follow-up time: PSI group (RSH≥20mm)
  Interventions: Procedure: Selective thoracolumbar fusion (STLF) surgery
- Non-PSI: we divided all patients into two groups according to their RSH in the final follow-up time: Non-PSI group (RSH≤20mm)
  Interventions: Procedure: Selective thoracolumbar fusion (STLF) surgery

INTERVENTIONS:
Procedure: Selective thoracolumbar fusion (STLF) surgery — Selective thoracolumbar fusion (STLF) surgery, is an established corrective surgical technique for spinal deformities with excellent outcomes over time

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is the most common three-dimensional deformity of the spine that is typically characterized by curvature in both the coronal and sagittal planes. Selective thoracolumbar fusion (STLF) surgery, is an established corrective surgical technique for spinal deformities with excellent outcomes over time1. The objective of AIS corrective surgery encompasses the rectification of coronal and spinal rotation deformities while concurrently restoring the sagittal profile. However, some scholars suggested that correcting the Cobb angle and rotation deformity of the main thoracic curve has been associated with a sacrifice of sagittal plane aligament. Some researchers observed that significant reduction of thoracic kyphosis (TK) after the coronal deformity was corrected in their study3-5. In addition, Li et al3 found that both lumbar lordosis(LL) and sacral slope (SS) decreased after STLF surgery in their study. The sagittal plane of the spine column should be considered a chain-like structure, one section's change, that leads to compensatory changes in other segments, enables the maintenance of balance6. In addition, some scoloars suggested that the decrease in thoracic kyphosis may caused by vertebral derotation in STLF surgery.

Postoperative shoulder imbalance (PSI) is a common complication that arises following STLF surgery, significantly impacting the appearance and satisfaction of patients8. The incidence of PSI varies within a range of 25% to 57%. It is imperative to identify the independent risk factors of PSI which can help in comprehending this phenomenon better and further aiding in deduction of the incidence rate. Although the research on the risk factors for PSI in AIS patients have been conducted for several years , no conclusively determination has been reached. Recently, scholars have been studying the relationship between the rotation of the thoracic spinal column and postoperative shoulder balance. Yagi et al.'s study10 has identified the preoperative rotation of the main thoracic apical vertebrae as a risk factor for PSI. Additionally, Masayoshi et al has reported on the relationship between the rotation of the proximal thoracic apical vertebrae and postoperative shoulder height disatance.

In summary, it can be hypothesized that the preoperative and changes of postoperative sagittal spinal parameters may impact the postoperative shoulder balance among AIS patients. However, there is a paucity of literature investigating the effect of sagittal spinal parameters on PSI after STLF surgery. Therefore, the purpose of this study is to examine the correlation between the preoperative and postoperative alterations of sagittal spinal parameters and PSI.

DETAILED DESCRIPTION:
PSI as a postoperative complication of Selective Thoracic-Lumbar Fusion (STLF) in AIS patients has been proven by numerous scholars to be an important factor affecting patients' satisfaction with the surgery and the mental health of adolescents, with an incidence rate of 25%-57%. Currently, most scholars' research on shoulder imbalance risk factors is mainly focused on coronal plane parameters and still remains highly controversial.In their study, Lee found that the preoperative Risser sign level of the PSI group was significantly higher than that of the non-PSI group during postoperative follow-up. Some domestic experts believe that the preoperative upper thoracic Cobb angle (PTC Cobb) and the ratio of preoperative upper thoracic to main thoracic curves (Pre PTC/MTC) have a certain predictive value for the occurrence of PSI after surgery. It has also been shown that the preoperative shoulder imbalance in the PSI group was significantly more severe than in the non-PSI group during the last follow-up. The preoperative presence of shoulder imbalance is of great significance in guiding the surgeon's choice of upper instrumented vertebra (UIV). Rose, Lenke, Qiu Yong, and others believe that different preoperative shoulder heights should lead to different choices of UIV. When the right shoulder is higher, it is recommended to fix the UIV at T4/T5, and when the preoperative shoulder height is already balanced, the UIV should be selected at T3 or T4. However, when the left shoulder is higher preoperatively, it should be fixed at the T2 level. Brooks, through a study of 648 AIS patients, found that the probability of PSI occurring after surgery in patients with UIV=T4 is the lowest compared to UIV=T2, T3, T5. Furthermore, incorrect correction of PTC and MTC by the surgeon can also lead to PSI in patients. Different researchers have given different answers on how to choose the appropriate PTC/MTC correction rate. Zhang and others believe that to prevent PSI in Lenke 1 patients after surgery, it is important to fully correct the upper thoracic curve and appropriately correct the main thoracic curve. In a study by John et al. on the risk factors for postoperative PSI in Lenke 1 and 2 patients, it was found that when the correction rate of the main thoracic curve was greater than 54% and the correction rate of the upper thoracic curve was less than 52%, 59% of the patients experienced PSI during the last follow-up. In a study by Ke et al., it was found that when the correction rate of the upper thoracic curve exceeded 55.3%, 88.4% of the individuals could maintain shoulder balance during the last follow-up, while when the correction rate of the main thoracic curve was greater than 56% and the correction rate of the upper thoracic curve was less than 55.3%, 66.3% of AIS patients would develop PSI at the last follow-up after surgery. Some experts believe that not only the position of the upper fixed vertebra affects the postoperative shoulder balance but also the choice of the lowest fixed vertebra affects the postoperative shoulder balance in AIS patients. To avoid the occurrence of PSI in AIS patients after surgery, Tatsuya Sate suggests that the lowest fixed vertebra should be selected at the lowest touchable vertebra (LTV) or the vertebra above LTV.

Although STLF can effectively improve the spinal deformity of AIS patients and has been used in clinical practice for many years, some scholars have found that while correcting the coronal imbalance of patients with this procedure, it often sacrifices the sagittal balance. The size of coronal and sagittal parameters in patients with spinal scoliosis can effectively assess the severity of spinal deformity. AIS, as a three-dimensional spinal deformity, has a correlation between sagittal and coronal deformities. Wu et al.'s study indicated that the main curve Cobb angle in AIS patients is related to sagittal parameters such as thoracic kyphosis (TK), lumbar lordosis (LL), and sacral slope (SS). Studies have shown that with the correction of the main curve, it may simultaneously lead to a decrease in sacral slope (SS) and an increase or decrease in thoracic kyphosis (TK). The sagittal structure of the spine is considered a chain-like structure, and when there is a change in any segment of the cervical, thoracic, lumbar spine, and pelvic segments, the remaining segments compensate to restore the sagittal alignment of the spine. Through the study of the shoulder joint and surrounding anatomy, it is known that the shoulder joint, spine, and clavicle are not directly connected but rely on soft tissues such as muscles and ligaments in between, and the support of the shoulder strap mainly relies on the rhomboid and trapezius muscles. The presence of the trapezius muscle allows the scapula to adhere closely to the chest wall, avoiding excessive elevation. When the strength of these muscles changes, the body may not be able to maintain shoulder balance. In recent years, it has been found that sagittal parameters of the spine, such as thoracic kyphosis and pelvic incidence angle, are related to the strength of the back muscles, such as the trapezius and rhomboid muscles. In addition, the magnitude of thoracic kyphosis (TK) may affect the rotation of the upper curve. Since the rotation axis of the spine is in front of the thoracic spine, when the thoracic kyphosis decreases, the distance between the thoracic vertebra and the spinal rotation axis is reduced, resulting in a simpler rotation of the thoracic vertebra in this segment. The final result may lead to an increase in the rotation degree of the upper curve. In recent years, Mitsuru Yagi proposed a new radiographic parameter, the Clavicle-Chest Cage Angle Difference (CCAD). Mitsuru Yagi found that the CCAD in patients with postoperative PSI group was significantly greater than that in the non-PSI group during preoperative, postoperative, and postoperative follow-up. Subsequent studies by Xiao et al. indicated that the preoperative CCAD can effectively predict whether AIS patients will develop PSI after surgery. Currently, the reasons for the occurrence of CCAD and how it affects postoperative shoulder balance in AIS remain inconclusive. Some scholars have proposed several possible reasons for CCAD leading to postoperative PSI in AIS patients: 1. The existence of residual CCAD after surgery may mean that there is residual rotational deformity in the upper curve of AIS patients after surgery. The residual rotational deformity of the upper curve may cause the elevation of the left shoulder, affecting the postoperative shoulder balance of the patients. 2. The residual rotation of the upper curve after surgery may lead to atrophy of the soft tissues connecting the shoulder joint, spine, causing atrophy of the shoulder joint, and eventually resulting in shoulder imbalance. The relationship between sagittal parameters of the spine and the strength of the soft tissues connecting the scapula, clavicle, and spine has been reported in previous studies. In conclusion, we hypothesize that the occurrence of postoperative PSI in AIS patients may be correlated with the preoperative and postoperative sagittal parameters of the patients Subject population

The subjects of this study sought medical treatment in the Department of Spinal Orthopedics, Southern Hospital, Southern Medical University, and referred to the "Clinical Practice

Diagnosis of adolescent idiopathic scoliosis using textbooks such as Orthopedics and Surgery, as well as imaging evidence

Adolescent idiopathic spine with protruding patients who require posterior selective thoracolumbar fusion surgery as determined by clinical physicians

Patients with scoliosis.

Diagnostic criteria:

The subjects of this study sought medical treatment in the Department of Spinal Orthopedics, Southern Hospital, Southern Medical University, and referred to the "Clinical Practice

Diagnosis of adolescent idiopathic scoliosis using textbooks such as Orthopedics and Surgery, as well as imaging evidence

Adolescent idiopathic spine with protruding patients who require posterior selective thoracolumbar fusion surgery as determined by clinical physicians

Patients with scoliosis.

Selection criteria:

1. Diagnosed as AIS upon admission;
2. The surgical age is 10-25 years old;
3. The surgical method is posterior selective thoracolumbar fusion;

The last reexamination was between January 2008 and May 2022;

5: AIS patients who need to collect complete imaging data before and after surgery;

5.3 Exclusion criteria:

Previous history of spinal trauma or spinal surgery;

6. Research methods and steps

This is a retrospective case-control study, with plans to collect the last follow-up in January 2008

AIS patients undergoing posterior selective thoracolumbar fusion surgery at the Spinal Orthopedics Department of Southern Hospital between May 2022

Preoperative and postoperative imaging data, and all collected imaging data will be used using IBM SPSS

25.0 (or higher) for statistical analysis without the need for additional visits, laboratory analysis, or routine analysis

Evaluation beyond clinical practice requirements. Doctors will determine treatment plans based on diagnostic and treatment standards. Researchers will investigate

Review the patient's medical history and laboratory reports to determine their eligibility based on inclusion and exclusion criteria. This research application

Exemption from being informed, as the samples and information involved in the study are sourced from clinical diagnosis and treatment records and specimens

The risk of the patient does not exceed the minimum risk, and exemption from knowing will not have adverse effects on the patient's rights or health

And if informed research is obtained, it will not be possible to conduct, and the privacy and personal identity information of the subjects will be protected.

Informed consent and enrollment

This study applies for exemption from informed consent forms, and subjects who meet all other inclusion/exclusion criteria are considered

For inclusion in this study.

Subject identification number

Each patient and clinical tissue sample is given a unique identification number based on the imaging findings at the last follow-up examination

Is the difference in shoulder height (RSH) greater than 20mm? Divide patients into PSI group (RSH ≥ 20mm) and Non PSI group

(RSH < 20mm). If the patient is in the Non PSI group and the enrollment order is 1, the identification number Non 01 will be given.

All research documents will use this identification number. This identification number does not contain any combination information that can identify the subject's identity.

Data source/data collection process

By collecting preoperative, postoperative, and follow-up imaging data from patients with AIS, this study aims to

data Case data, detailed data of relevant imaging parameters, and identification numbers are uniformly recorded by the researchers in the experiment

In the record table.

Data collection steps

Record demographic data: age, gender;

Collect preoperative and postoperative imaging parameters of patients included in this study; 7. Study Termination/Suspension Criteria

The applicant has the right to terminate/suspend this study. Applicants must be notified before terminating/suspending a clinical study

Researchers, ethics committees, and relevant regulatory authorities, and provide reasons. After early termination/suspension of the study, re

New research must be reviewed and approved by the ethics committee;

Termination/suspension requested by the Ethics Committee.

Provisions for ending clinical research.

All preoperative and postoperative imaging data of included patients have been collected.

data management

1 Data Management

1. Researchers must ensure that the data is true, complete, and accurate;
2. When making any corrections to the research records, only underline and annotate the revised data, explain the reasons, and have the research

   Please sign and indicate the date, and do not erase or overwrite the original record;
3. The laboratory inspection items are complete.

Data recording and file storage

The relevant subject data on the case report form should be recorded in the subject coding format, and subjects can only use the

Identification of the subject's code or initials.

This study uses Microsoft Office for data management, and the verification from data entry to source data requires

Seek answers to questions about quality control data, and finally, after confirming the operation of data locking and exporting, and confirming that there are no doubts about the data,

All parties sign the database locking application form, and the data administrator will lock the database. After the database is locked,

Export the analysis database by the data administrator and submit it to the statisticians for statistical analysis. Locked data is not available

After further editing and database locking, any issues found can be corrected in the statistical analysis program after confirmation.

statistical analysis

Sample size determination

This study is a retrospective case study aimed at exploring the risk factors for shoulder imbalance in AIS patients after surgery

In a controlled study, the total sample size for current research on disease risk factors is 5-10% of the required number of factors to be explored

Therefore, this study plans to include 100 patients who meet the inclusion and exclusion criteria.

statistical method

The analysis content includes case distribution, demographic data, and relevant imaging data that needs to be collected for this study.

Statistical software and general requirements: All statistical analysis shall be completed using IBM SPSS 25.0 (or higher version).

Measurement data is described using mean, standard deviation, median, maximum, and minimum values

Count data using frequency and percentage descriptions

Research management

Comply with relevant regulatory requirements

1. Researchers should use standard operating procedures to conduct quality control and quality assurance systems for clinical studies;
2. The original data must comply with relevant regulatory requirements;
3. The laboratory inspection results must be accurate and reliable;
4. All observations and findings used should be verified to ensure the reliability of the data;
5. Establish a complete research organization and clarify the responsibilities of personnel at all levels;
6. The main researchers are responsible for comprehensive quality control and carry out the responsibilities of personnel at all levels;
7. The main researcher is responsible for designing the research protocol and informed consent form. After the study is completed, the main researcher

   Write a research summary report;
8. The designated researcher is responsible for developing research implementation rules and SOPs for use in the study;
9. Before the study, the research group organizes a learning plan for all participants, and all participants must go through the

   GCP training;
10. Physicians and nurses participating in the study must strictly abide by the protocol regulations, follow the procedures, and are not allowed to change at will

    Change;
11. The designated statistician is responsible for the comprehensive statistical processing of the data.

Protecting the privacy of subjects

All data of the subjects during the study period will be entered into a computer for confidential storage and analysis, if necessary

The shutdown organization may review the records to verify the authenticity, accuracy, and completeness of the data, and study the obtained information

It may also be published in academic journals, but the names of the participants will not be disclosed and their privacy will be kept confidential.

Take additional preventive measures to ensure the confidentiality of documents and prevent the identification of subjects based on genetic data

Identity. However, in special circumstances, some individuals may see the genetic data and individuals of a certain subject

Identification code. For example, in the event of medical emergency, the sponsor, their representative doctor, or researcher is aware that

Subject identification code and access to the subject's genetic data. In addition, relevant regulatory agencies require

Access relevant files.

The problems that occurred during the research and their handling measures 1) Revision of the plan: After approval by the Ethics Committee, if this plan needs to be revised, a "Plan Revision

Order instructions "and signed by the main researcher;

2) After the plan is revised, it must be submitted to the Ethics Committee for review and approval before implementation;

3) No participant in the study shall violate the protocol.

Quality Control and Quality Assurance

Quality assurance:

A cooperation agreement between the applicant and the person entrusted by the applicant to be responsible for all or part of the responsibilities and tasks related to this study

Each department (including CRO, SMO, statistical unit, clinical center, etc.) should establish their own quality assurance bodies

Department, fulfill their respective responsibilities, strictly follow the clinical research protocol, and adopt corresponding standard operating procedures,

To ensure the implementation of clinical research quality control and quality assurance system.

Quality assurance of clinical research process

Before initiation, researchers should receive training on the research protocol to enable them to understand the clinical research protocol and its

There is a thorough understanding and understanding of the specific connotations of each indicator. Quality control personnel should verify the basic conditions of clinical research,

Ensure that the clinical research conditions meet the protocol requirements. During the research process, researchers should follow the institutional SOP and research

The plan requires careful execution of clinical procedures and other work, and truthful, timely, complete, and standardized recording.

Quality control personnel conduct quality checks on the research process and corresponding original records. After the study is completed, the study form

Organize the corresponding project documents, verify them by quality control personnel, and archive and save them. Quality Assurance of Clinical Research Units

The department conducts feasibility checks on the research conducted. Notify researchers promptly when non conformities are found

Make corrections with the unit leader and track the progress of the corrections.

ELIGIBILITY:
Inclusion Criteria:

- (i): diagnosed with Lenke 1/2 AIS;(ii).underwent the selective thoracolumbar fusion;

Exclusion Criteria:

* (i).were diagnosed with other types scoliosis(eg, congenital, neuromuscular) (ii).lacked preoperatively, immediately postoperatively, or follow-up time radiographic data.

Ages: 10 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The subjects of this study sought medical treatment in the Department of Spinal Orthopedics, Southern Hospital, Southern Medical University, and referred to the "Clinical Practice Diagnosis of adolescent idiopathic scoliosis using textbooks such as Orthopedics and Surgery, as well as imaging evidence
  Adolescent idiopathic spine with protruding patients who require posterior selective thoracolumbar fusion surgery as determined by clinical physicians
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
RSH | baseline, immediately after, and at least 2 years after surgery.
  RSH was measured as the linear distance between the horizontal reference lines, passing through the soft tissue shadow of the shoulder directly above the acromial clavicular joint of each shoulder.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China